CLINICAL TRIAL: NCT02020551
Title: Lidocaine 10% Spray Reduces Pain During Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Açmaz, MD, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: kerhGA
Record Dates: First submitted 2013-12-11; First posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Pain
Keywords: Scores During IUD insertion.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline spray application (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo
- lidocaine spray application (Experimental): 2 puff lidocaine spray applicated before IUD insertion
  Interventions: Drug: Lidocaine Spray

INTERVENTIONS:
Drug: Lidocaine Spray
  Arms: lidocaine spray application
Drug: Placebo
  Arms: saline spray application

SUMMARY:
Pain during intrauterine device (IUD) insertion can be a barrier to initiation. Misoprostol and nonsteroidal drugs have found to be ineffective by clinical trials.Investigators tested whether intracervical 2% lidocaine gel decreased insertion pain compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Age >18 Not pregnant Smear negative

Exclusion Criteria:

Chronic pelvic pain Pregnancy Uterine anomaly Fibroid Acute cervicitis Pelvic inflammatory disease Cervical stenosis

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pain | 3 months
  10 cm VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Education and Research Hospital of Medicine, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Aksoy H, Aksoy U, Ozyurt S, Acmaz G, Babayigit M. Lidocaine 10% spray to the cervix reduces pain during intrauterine device insertion: a double-blind randomised controlled trial. J Fam Plann Reprod Health Care. 2016 Apr;42(2):83-7. doi: 10.1136/jfprhc-2014-100917. Epub 2015 Mar 10. PMID 25759418